CLINICAL TRIAL: NCT04439552
Title: Neuroplasticity of Pain Pathways and Corneal Afferent Regeneration Following Corneal Crosslinking (CXL) in Keratoconus
Brief Title: fMRI and IVCM Cornea Microscopy of CXL in Keratoconus
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Eric Moulton, Assistant Professor of Anesthesia, Boston Children's Hospital
Other Study IDs: IRB-P00035185
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Pain, Postoperative; Pain, Chronic; Pain, Acute; Surgical Injury; Surgical Wound; Cornea Injury; Cornea; Keratoconus
Keywords: fMRI; Corneal Microscopy; IVCM; Neuroimaging
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain; Acute Pain; Intraoperative Complications; Surgical Wound; Corneal Injuries; Corneal Diseases; Keratoconus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CXL group: Patients who are about to undergo a corneal cross-linking (CXL) surgery to treat keratoconus.
- Control group: Healthy volunteers age and sex matched to the CXL group.

SUMMARY:
Evaluation of neuroplasticity of pain pathways and corneal afferent nerve regeneration following corneal crosslinking (CXL) in keratoconus patients using fMRI and corneal In Vivo Confocal Microscopy (IVCM).

DETAILED DESCRIPTION:
Our long-term goal is to evaluate the transition from acute to chronic pain that sometimes occurs following CXL in keratoconus patients. This study will determine whether these changes can be structurally and functionally quantified using functional neuroimaging and in vivo corneal microscopy (IVCM), and whether they can be predicted based on predisposing biological and psychological factors. Our central hypothesis is that CXL produces acute pain through activation of trigeminal afferents, and that post-operative chronic pain outcomes are related to neuroplastic changes in trigeminal circuitry, corneal afferent regeneration, and psychological factors.

ELIGIBILITY:
Inclusion Criteria:

CXL Group

* Age 8-35 years
* Clinical diagnosis of keratoconus and seeking CXL treatment
* English speaking ability sufficient to comprehend consent with parental assistance
* MRI compatible
* Ability to lie still for an MRI session (60 minutes)

Control Group

* Age 8-35 years
* No diagnosis of keratoconus
* English speaking ability sufficient to comprehend consent with parental assistance
* MRI compatible
* Ability to lie still for an MRI session (60 minutes)

Exclusion Criteria (Both Groups):

* Claustrophobic
* Weight > 285 lbs (weight limit of the MRI table)
* Significant medical history, including:

Current DSM-IV-TR axis I psychiatric disorders. Chronic pain Significant head injury Seizures Brain tumor Cerebrovascular accident Neurological disease aside from migraine HIV-AIDs Prescription medication strongly implicated in causing dry eyes

* Magnetic implants or metal-containing tattoos on their chest or above
* Pregnancy
* History of contact lens wear
* Any allergic response to a numbing eyedrop in the past

Ages: 8 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The population under study are patients with keratoconus who are undergoing a corneal cross-linking (CXL) procedure. Keratoconus is an eye condition where the cornea progressively develops abnormally into a cone shape, which can lead to distorted vision and irreversible vision loss The CXL procedure is designed to restore and maintain the shape of the cornea to avoid these complications.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-10-04 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Neural activity related to pain. | 1 year
  Pain-related brain activation measured with fMRI.
Corneal nerve morphology. | 1 year
  Afferent nerve fiber morphology measured with IVCM.

CONTACTS AND LOCATIONS:
Overall Officials: Eric A Moulton, OD PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication, until 5 years after.
Access Criteria: Direct request to study personnel via email, letter, phone, or in-person communication. Information will be shared with requesting parties for the purposes of expanding on this research or re-analysis. Neuroimaging data and corneal microscopy data will be shared via secure digital electronic transfer.

REFERENCES:
- [Background] Belmonte C, Acosta MC, Merayo-Lloves J, Gallar J. What Causes Eye Pain? Curr Ophthalmol Rep. 2015;3(2):111-121. doi: 10.1007/s40135-015-0073-9. PMID 26000205
- [Background] Borsook D, Youssef AM, Simons L, Elman I, Eccleston C. When pain gets stuck: the evolution of pain chronification and treatment resistance. Pain. 2018 Dec;159(12):2421-2436. doi: 10.1097/j.pain.0000000000001401. PMID 30234696
- [Background] Cruzat A, Qazi Y, Hamrah P. In Vivo Confocal Microscopy of Corneal Nerves in Health and Disease. Ocul Surf. 2017 Jan;15(1):15-47. doi: 10.1016/j.jtos.2016.09.004. Epub 2016 Oct 19. PMID 27771327
- [Background] Downie LE, Naranjo Golborne C, Chen M, Ho N, Hoac C, Liyanapathirana D, Luo C, Wu RB, Chinnery HR. Recovery of the sub-basal nerve plexus and superficial nerve terminals after corneal epithelial injury in mice. Exp Eye Res. 2018 Jun;171:92-100. doi: 10.1016/j.exer.2018.03.012. Epub 2018 Mar 14. PMID 29550279
- [Background] Ghanem VC, Ghanem RC, de Oliveira R. Postoperative pain after corneal collagen cross-linking. Cornea. 2013 Jan;32(1):20-4. doi: 10.1097/ICO.0b013e31824d6fe3. PMID 22547128
- [Background] Hruschak V, Cochran G. Psychosocial predictors in the transition from acute to chronic pain: a systematic review. Psychol Health Med. 2018 Dec;23(10):1151-1167. doi: 10.1080/13548506.2018.1446097. Epub 2018 Feb 28. PMID 29490476
- [Background] Hasenbring MI, Chehadi O, Titze C, Kreddig N. Fear and anxiety in the transition from acute to chronic pain: there is evidence for endurance besides avoidance. Pain Manag. 2014;4(5):363-74. doi: 10.2217/pmt.14.36. PMID 25350076
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Kennedy RH, Bourne WM, Dyer JA. A 48-year clinical and epidemiologic study of keratoconus. Am J Ophthalmol. 1986 Mar 15;101(3):267-73. doi: 10.1016/0002-9394(86)90817-2. PMID 3513592
- [Background] Kinard KI, Smith AG, Singleton JR, Lessard MK, Katz BJ, Warner JE, Crum AV, Mifflin MD, Brennan KC, Digre KB. Chronic migraine is associated with reduced corneal nerve fiber density and symptoms of dry eye. Headache. 2015 Apr;55(4):543-9. doi: 10.1111/head.12547. Epub 2015 Mar 31. PMID 25828778
- [Background] Larbig W, Andoh J, Huse E, Stahl-Corino D, Montoya P, Seltzer Z, Flor H. Pre- and postoperative predictors of phantom limb pain. Neurosci Lett. 2019 May 29;702:44-50. doi: 10.1016/j.neulet.2018.11.044. Epub 2018 Nov 29. PMID 30503915
- [Background] Moulton EA, Becerra L, Borsook D. An fMRI case report of photophobia: activation of the trigeminal nociceptive pathway. Pain. 2009 Oct;145(3):358-363. doi: 10.1016/j.pain.2009.07.018. Epub 2009 Aug 11. PMID 19674842
- [Background] Moulton EA, Borsook D. C-Fiber Assays in the Cornea vs. Skin. Brain Sci. 2019 Nov 12;9(11):320. doi: 10.3390/brainsci9110320. PMID 31718074
- [Background] Rosenthal P, Borsook D, Moulton EA. Oculofacial Pain: Corneal Nerve Damage Leading to Pain Beyond the Eye. Invest Ophthalmol Vis Sci. 2016 Oct 1;57(13):5285-5287. doi: 10.1167/iovs.16-20557. PMID 27723896
- [Background] Schiffman RM, Christianson MD, Jacobsen G, Hirsch JD, Reis BL. Reliability and validity of the Ocular Surface Disease Index. Arch Ophthalmol. 2000 May;118(5):615-21. doi: 10.1001/archopht.118.5.615. PMID 10815152
- [Background] Simone DA, Nolano M, Johnson T, Wendelschafer-Crabb G, Kennedy WR. Intradermal injection of capsaicin in humans produces degeneration and subsequent reinnervation of epidermal nerve fibers: correlation with sensory function. J Neurosci. 1998 Nov 1;18(21):8947-59. doi: 10.1523/JNEUROSCI.18-21-08947.1998. PMID 9787000
- [Background] Sjoberg J, Kanje M. The initial period of peripheral nerve regeneration and the importance of the local environment for the conditioning lesion effect. Brain Res. 1990 Oct 8;529(1-2):79-84. doi: 10.1016/0006-8993(90)90812-p. PMID 2282506
- [Background] Tervo K, Latvala TM, Tervo TM. Recovery of corneal innervation following photorefractive keratoablation. Arch Ophthalmol. 1994 Nov;112(11):1466-70. doi: 10.1001/archopht.1994.01090230080025. PMID 7980137
- [Background] Pondelis NJ, Moulton EA. Supraspinal Mechanisms Underlying Ocular Pain. Front Med (Lausanne). 2022 Feb 8;8:768649. doi: 10.3389/fmed.2021.768649. eCollection 2021. PMID 35211480
- [Background] van der Valk Bouman ES, Pump H, Borsook D, Severinsky B, Wisse RP, Saeed HN, Moulton EA. Pain mechanisms and management in corneal cross-linking: a review. BMJ Open Ophthalmol. 2021 Nov 29;6(1):e000878. doi: 10.1136/bmjophth-2021-000878. eCollection 2021. PMID 34901466
- [Background] Dieckmann G, Borsook D, Moulton E. Neuropathic corneal pain and dry eye: a continuum of nociception. Br J Ophthalmol. 2022 Aug;106(8):1039-1043. doi: 10.1136/bjophthalmol-2020-318469. Epub 2021 Apr 30. PMID 33931393